CLINICAL TRIAL: NCT01317238
Title: An Open-label, Single Arm, Phase III Clinical Study to Evaluate the Efficacy and Safety of CJ Smallpox Vaccine in Previously Vaccinated Healthy Volunteers
Brief Title: Safety and Efficacy of CJ Smallpox Vaccine in Previously Vaccinated Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CJ_SPX_303; CJ corporation
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Smallpox
Keywords: Smallpox vaccine efficacy
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CJ Vaccination arm (Experimental): healthy vaccinia-experienced volunteers who received CJ smallpox vaccine
  Interventions: Drug: smallpox vaccine CJ-50300

INTERVENTIONS:
Drug: smallpox vaccine CJ-50300 — Conventional CJ-50300 2.5 x 100000 pfu/dose vaccination
  Other Names: CJ-53300

SUMMARY:
The currently available stock of smallpox vaccine would be insufficient in the face of an incident of smallpox attack. Thus, new manufacturing methods for smallpox vaccine are urgently needed because previous manufacturing methods using calf lymph are no longer acceptable in the view of current standards. Recently, CJ corporation in Republic of Korea has developed cell-culture derived smallpox vaccine (CJ-50300) which was manufactured by infecting MRC-5 cells. The aim of this clinical trial were to assess safety, reactogenicity, and immunogenicity of CJ-50300 in previously vaccinated healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean male and female subjects below 60 years of age and born before 1979.
2. subjects who have been vaccinated wiht smallpox vaccines
3. Willing to participate and have signed the informed consent form
4. In good general health, without clinically skin diseases history, physical examination or laboratory test results
5. Hematocrit > 33% for women; > 38% for men
6. White cell count 3,300-12,000/mm3
7. Total lymphocyte count > 800 cells/mm3

Exclusion Criteria:

1. Subjects who were born after 1980
2. Diseases or conditions that cause immunodeficiency (For examples; HIV AIDS, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, history of transplantation, therapy with alkylating agents, antimetabolites, radiation, or oral or parenteral corticosteroids, basal cell carcinoma, liver cirrhosis or advanced liver disease).
3. In close physical contact (household or at work) with an individual who has the diseases or conditions that cause immunodeficiency
4. History or present of eczema or atopic dermatitis
5. Allergy or sensitivity to any known components of vaccine or other medicines
6. In close physical contact (household or at work) with an individual who has acute or chronic skin conditions such as dermatitis, exfoliative dermatitis
7. Subjects who have taken corticosteroid within 3 months of vaccination or who are taking oral or parenteral corticosteroid.
8. Subjects who have been taken immunosuppressive therapy including interferon within 3 months of vaccination or are taking immunosuppressive therapy.
9. subjects who are planning for blood donations
10. Autoimmune disease such as lupus erythematosus
11. Subjects who work in medical institution
12. Household contacts with women who are pregnant or breast-feeding
13. Female subjects who are pregnant or breast-feeding and have positive result by serum pregnancy test or urine pregnancy test, or do not using approved contraceptives such as sterilization, contraceptive ring injectable, combined oral contraceptive pills and barrier contraceptive, combined hormone-based therapy, contraceptive cream, contraceptive jelly, diaphragm or condoms
14. Subjects household member < 1 year old or work with children < 1 year old
15. Subjects with a known history of Cardiac disease or have three or more of the following risk factors: hyperpiesia, obesity, hyperlipidemia, glucosuria, sclerosis, cerebral arteriosclerosis
16. Receipt of immunoglobulin or vaccine within 4 weeks of vaccination
17. Subjects who are allergic to latex, inflammatory opthalmic disease, or taking antiviral agents.
18. Receipt of investigational research agents within 4 months of vaccination
19. HBsAg seropositive
20. HCV antibody seropositive
21. HIV seropositive
22. Subjects having fever (oral temperature > 38℃) or severe nutrition disorder
23. Blood donation within 3 months since screening visit
24. Subject who are not suitable to participate in study according to investigator's judgement

Ages: 32 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pocket formation | 7-9 day
Adverse reactions | 0-28 days

SECONDARY OUTCOMES:
Antibody response | 14 or 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea